CLINICAL TRIAL: NCT05655572
Title: Comparison Between Action Observation Therapy and Functional Training on Balance, Mobility and Cognition in Diplegic Cerebral Palsy
Brief Title: Comparison Between AOT and Functional Training on Balance, Mobility and Cognition in Diplegic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Aizaz Ullah Khan
Record Dates: First submitted 2022-12-09; First posted 2022-12-19 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Diplegic Cerebral Palsy
Keywords: Action observation therapy (AOT); Cerebral Palsy (CP)
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Action Observation therapy (Experimental): This group will perform exercises in stages. First stage consists of movements to improve balance in sitting position with exercises upright the pelvis, move weight forward, move weight to the left and right and rotate right and left. Second stage consist of sit to stand movements with exercises upright the pelvis in sitting position, move weight forward from a sitting position and stand up from a sitting position. Third stage consist of standing movements to improve balance with exercises move weight right and left, forward weight shift with right foot and left foot (lateral view) and forward weight shift with right foot and left foot (front view). Fourth stage consist of walking side ways to left and then towards right. Therapist will perform these tasks and video will be made which will play in front of patients.
  Interventions: Other: Action Observation Theraoy
- Functional Training Group (Active Comparator): participants including in this group will perform the tasks including lying to sitting position, moving in the sitting posture, sitting and standing up, posture training for learning a normal gait pattern, weight bearing and weight movement training in the straight posture, walking training on the flat floor, and stair walking
  Interventions: Other: Functional Training

INTERVENTIONS:
Other: Action Observation Theraoy — After initial baseline assessment patients allocated in AOT group will undergo treatment protocol of 6 weeks having 4 stages of duration 1.5 weeks each performed 3 days per week. . Assessment will be perform at baseline after 2, 4 and 6 weeks
  Arms: Action Observation therapy
Other: Functional Training — after baseline assessment participants including in this group will perform the tasks for 6 weeks (3 days per week) s and after that again assessment will be made for examining the improvements.Assessment will be perform at baseline after 2 ,4 and 6 weeks
  Arms: Functional Training Group

SUMMARY:
The aim of the study is to find out the effects of Action observation therapy as compared to the traditional physiotherapy in diplegic spastic cerebral palsy patients. We will check the effects on balance mobility and cognition of patients.

DETAILED DESCRIPTION:
A study conducted in 2020 on diplegic CP patients. The action observation training group repeatedly practiced the action with their motor skills, while the control group practiced conventional physical therapy. Results suggest that action observation training is both feasible and beneficial for improving spasticity, gross motor function, and balance in children with spastic diplegia cerebral palsy.

One of the researcher evaluated the evidence of using Action Observation Therapy in the rehabilitation of children with Cerebral Palsy. It was Systematic review with meta-analysis. No evidence of benefit had been found to draw a firm conclusion regarding the effectiveness of action observation therapy in the rehabilitation of children with cerebral palsy due to limitations in methodological quality and variations between studies.

Some also, investigated the effects of VR-based intervention by means of active videogame on self-concept, balance, motor performance and adaptive success in children with CP. They concluded that VR-based intervention might interfere with the way children with CP perceive themselves, apart from improve their balance, motor performance and adaptive success. Thus VR-based intervention is a potential tool to assist rehabilitation professionals to improve these aspects of children's health condition.

Similarly, A study concluded that Action observation therapy is beneficial in rehabilitation of neurological and musculoskeletal conditions. A study concluded that action observation along with gait training provides greater benefits for gait and cognitive performance in elderly with MCI. According to a scientist action observation therapy is effective and feasible for functional mobility in rehabilitation processes. A researcher in his study action observation therapy is more effective in improving upper limb movements and functions.

There are various studies on movement observation training but most of them are related to restoring the upper limb function of stroke and cerebral palsy patients, and studies on the mobility, cognition, and balance in cerebral palsy for movement observation training are sparse so this study will contribute in examining improvements in rehabilitation of children with diplegic cerebral palsy by demonstrating the effects of action observation training and conventional therapy for the treatment of mobility, cognition, and balance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Diaplegic Spastic CP between the age of 5 to 11 years.
* Able to follow the researcher's instruction.
* GMFCS (gross motor function classification system) level I-III
* Children with a modified ashworth scale (MAS) of ≤ 3.

Exclusion Criteria:

* Unable to walk
* Children with severe co-morbidities like musculoskeletal deformities, spina bifida and other types of Cerebral Palsy.
* With visual impairment and visual field defects

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Gross motor function measure | 6 weeks
  Changes form the baseline Gross Motor Function measure (GMFM) is the valid and standard observational instrument to measure change in gross motor function in CP children. It consists of 66 items with 5 dimensions. These dimensions are the major motor functions i.e. supine/rolling, sitting, crawling/kneeling, standing and walking/running/jumping. Each task is rated according to the scoring guidelines i.e. higher score indicated better gross motor function. Each GMFM item is graded on 4-point scale i.e. 0 for unable to initiate the task, 1 for able to initiate the task, 2 for able to perform the task partially and 3 for able to perform the task completely
Pediatric Balance Scale (PBS) | 6 weeks
  Changes from the baseline Pediatric Balance Scale (PBS) is a modified form of Berg Balance Scale (BSS) which was developed for balance measurement in CP child. It can be performed without specialized equipment and can be easily administered. It including 14 items with 5-level grading to assess the functional activities that child must safely and independently form at home, community, activities including sitting balance, sit to stand/stand to sit, transfer, stepping, reaching forward, reaching to floor, turning and stepping on and off at elevated surface. Each activity is rated according to scale from 0 to 4 i.e. 0 for unable to perform and 4 for able to perform without difficulty.
Timed 10 meter walk test | 6 weeks
  Changes from baseline Timed 10 meter walk test was used to measure the gait ability and speed. The acceleration area 2.5m and deceleration area 2.5m were marked on the ground as start and end point for the test. Participants were asked to walk for 15 minutes on comfortable flat floor at a comfortable speed and then record the walking speed through stopwatch over 10 m between these point
Mini-mental state pediatric examination (MMSPE) | 6 weeks
  Changes from baseline Mini-mental state pediatric examination (MMSPE) is a cognitive screening task and scoring system for 3 to 14 years old child. It represented 11 questions involving five basic cognitive abilities i.e. attention-concentration, orientation, registration, recall and language and constructive ability. (22) The possible score range is from 0 to 37, from which 17 or lower score indicating as moderate to severe cognitive impairment of children.

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Bashir, MSNMPT, Principal Investigator — Riphah International University
Locations (1):
- Saidu Group of Teaching Hospital Swat, Swāt, Khyberpakhtunkhuwa, Pakistan

IPD SHARING:
Plan to Share IPD: No